CLINICAL TRIAL: NCT06603194
Title: BECOME Study: Comparative Efficacy of Bovine and Marine Collagen Versus Placebo on Skin, Hair, Nails and Whole Body Health Markers
Brief Title: Benefit of Bovine or Marine Collagen Vs. Placebo on Skin, Hair, Nails and Whole Body Health in Healthy Adults
Acronym: BECOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ancient + Brave (Industry)
Collaborators: Princeton Consumer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AABVIV1C
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Skin Laxity; Hair Thinning; Nails
Keywords: Collagen; Skin health; Skin density
MeSH Terms: conditions — Cutis Laxa; Alopecia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bovine Collagen (Active Comparator): 10g powder format taken daily for duration of the study.
  Interventions: Dietary Supplement: Bovine or Marine Collagen
- Marine Collagen (Active Comparator): 10g powder format taken daily for duration of the study.
  Interventions: Dietary Supplement: Bovine or Marine Collagen
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Bovine or Marine Collagen

INTERVENTIONS:
Dietary Supplement: Bovine or Marine Collagen — Bovine or Marine Collagen

SUMMARY:
The BECOME Study (Bovine and Marine Collagen Efficacy for Skin, Hair, Nails and Whole Body Health Markers Evaluation) is a randomized controlled trial designed to compare the effects of bovine and marine collagen supplements versus a placebo on skin, hair, nails and whole body health markers. The trial aims to determine the most efficacious collagen source for improving health outcomes and to establish if both types of collagen are equally effective. Participants will be assessed on various health parameters, including skin elasticity, joint health, digestive health, and overall well-being, over a specified period.

ELIGIBILITY:
Inclusion Criteria:

Females aged 35-55 years. Participants must be comfortable with bovine or marine collagen (non-vegan/vegetarian).

Must provide informed consent and be willing to comply with study requirements.

Exclusion Criteria:

Pregnant or breastfeeding women. History of chronic skin conditions (e.g., eczema, psoriasis) that might interfere with study outcomes.

Any active skin infections or severe acne. Currently taking collagen supplements or have taken them within the last 6 months.

Use of medications or topical agents that can affect skin, hair, nails, or gastrointestinal health (e.g., corticosteroids, retinoids).

Excessive alcohol consumption or current smokers. Regular use of sunbeds. Recent cosmetic procedures (e.g., Botox, fillers, chemical peels, laser treatments) on skin, hair, or nails within the last 3 months.

Any condition or situation that, in the opinion of the investigator, may interfere with the participant's ability to comply with the study requirements or give informed consent.

Poor adherence to previous study protocols

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2024-11-25 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in nail strength and growth | Baseline, week 6 and week 12
  Assessment of nail strength and growth will be assessed by self-perception questionnaire
Change in skin elasticity | Baseline, week 6 and week 12
  Changes in skin elasticity will be measured by a cutometer
Change in hair thickness and strength | Baseline, week 6 and week 12
  Strength and breakage of hair will be assessed by self perception questionnaire
Change in skin wrinkles | Baseline, week 6 and week 12
  Measurement of the reduction in skin wrinkles using Profilometer
Change in perceived skin health | Baseline, week 6 and week 12
  Changes in perceived skin health assessed by self perception questionnaire
Change in skin wrinkles by visual assessment | Baseline, week 6 and week 12
  Change in skin wrinkles will be performed by visual assessment by a dermatologist
Changes in skin pigmentation | Baseline, week 6 and week 12
  Changes in skin pigmentation will be assessed by Chromameter
Changes in skin hydration | Baseline, week 6 and week 12
  Changes in skin hydration will be assessed by a Corneometer

SECONDARY OUTCOMES:
Digestive Quality of Life (DQDL) Assessment | Baseline, week 6 and week 12
  Participants will complete a Digestive Quality of Life (DQDL) Assessment to evaluate the digestive health benefits
Subjective Perception Questionnaire | Baseline, week 6 and week 12
  Subjective Perception Questionnaire (SPQ) for Whole Body Health to capture participants' self-reported perceptions of their overall health and well-being

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Macciochi, PhD, Principal Investigator — jenna@ancientandbrave.earth; Becky Clarke, Study Director — Princeton Consumer Research
Locations (1):
- Princeton Consumer Research, 8 Richmond Road, Dukes Park, Chelmsford, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided